CLINICAL TRIAL: NCT05537324
Title: Effects of a Single Dose of Brazil Nuts on Blood Lipids. A Randomised Controlled Trial.
Brief Title: Effects of a Single Dose of Brazil Nuts on Blood Lipids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skogli Health and Rehabilitation Center (Other)
Responsible Party: Principal Investigator, Allan Fjelmberg, Medical director, Skogli Health and Rehabilitation Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Skonøtt
Record Dates: First submitted 2022-08-04; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Cholesterol Level, High
Keywords: Blood lipids, Brazil nut, coconut
MeSH Terms: conditions — Hypercholesterolemia | interventions — 2S albumin, brazil nut

STUDY DESIGN:
Intervention Model Description: This study was a non-blinded randomized controlled trial, where participants were requited and enrolled to the study / intervention continuously over about two years. Half of the participants (26) in the experimental group and half of the participants in the control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brazil nut (Experimental): 50g Brazil nuts
  Interventions: Other: Brazil nut
- Coconut (Other): 46g Coconut flakes
  Interventions: Other: Coconut

INTERVENTIONS:
Other: Brazil nut — Blood lipids are measured at baseline and 3h, 6h, 24h, 7d and 14d after ingestion of 50g Brazil nuts
  Arms: Brazil nut
Other: Coconut — Blood lipids are measured at baseline and 3h, 6h, 24h, 7d and 14d after ingestion of 46g coconut flakes
  Arms: Coconut

SUMMARY:
Several studies have shown that regular intake of nuts may improve blood lipids. However, few studies have investigated the effects on blood lipids after a single intake of nuts. The present study was conducted in order to evaluate the acute effects of a single intake of Brazil nuts on blood lipids.

The study was a non-blinded randomized controlled study with 52 participants, 26 participants in both the Brazil nut group and in the control group. Blood tests were taken at baseline and 3h, 6h, 24h, 7d and 14d after ingestion of either 50g Brazil nuts or an isocaloric amount of coconut flakes. We then conducted an unpaired t-test in order to compare changes in blood lipids between the two groups. P-values < 0.05 were considered statistically significant

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated in a rehabilitation program over three weeks at a rehabilitation center. Participants were at the rehabilitation center due to rheumatic diseases or chronic pain conditions / fibromyalgia.

Exclusion Criteria:

* Food allergy, lactose intolerance, celiac disease, mild illness for the last 3 weeks (infections or inflammatory conditions), serious illness (eg. heart attack) or undergone surgery during the previous 3 months, intake of Brazil four weeks prior study enrollment, using cholesterol-lowering or blood-thinning drugs, planning to eat more than one meal in other places than the rehabilitation center during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Changes in total cholesterol, LDL cholesterol and HDL cholesterol (mmol/l) | Blood tests are measured at baseline, 3 hours, 6 hours, 24 hours, 7 days and 14 days after intervention
  Changes in total cholesterol, LDL cholesterol and HDL cholesterol (mmol/l) between the experimental group and the control group at specific times after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Allan Fjelmberg, MD, MPH, Principal Investigator — Skogli Health and Rehabilitation Center
Locations (1):
- Skogli Health and Rehabilitation Center, Lillehammer, Innlandet, Norway

IPD SHARING:
Plan to Share IPD: No